CLINICAL TRIAL: NCT05096767
Title: Descriptors of Neuropathic Spinal Pain and Their Relations With Functional Status in Ankylosing Spondylitis Patients
Brief Title: Neuropathic Spinal Pain Descriptors in Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Taciser Kaya, Professor, MD, Bozyaka Training and Research Hospital
Other Study IDs: 355148EA
Record Dates: First submitted 2021-10-12; First posted 2021-10-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Surveys and Questionnaires; Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: questionnaires and inventories — questionnaires and inventories related to primary end secondary outcomes will be applied and physical examination will be performed

SUMMARY:
The investigators have aimed to explore and interpret the neuropathic pain (NP) descriptors of spinal pain in patients with ankylosing spondylitis (AS). For this purpose they have attempted to initiate a prospective, cross-sectional study with AS patients.

DETAILED DESCRIPTION:
NP descriptors have been investigated in several pain syndromes such as post-herpetic neuralgia, post-surgical nerve trauma, peripheral diabetic neuropathy and low back pain. But there is no study examining descriptors of inflammatory spinal pain with or without neuropathic characteristics seen in AS. To date, only one study reported distribution of sensory descriptors in neuropathic and non-neuropathic pain (nonNP) in AS patients, but in this paper the painful region was not specified and the results related to sensory descriptors were not discussed. Therefore, investigators have aimed to explore and interpret the sensory descriptors of inflammatory spinal pain in patients with AS. For this purpose investigators have attempted to initiate a study investigating whether sensory descriptors in neuropathic pain (NP) are differ from those seen in non-neuropathic pain (nonNP).

The aims of this study are;

1. To determine NP descriptors that associated with spinal pain in ankylosing spondylitis patients
2. To compare the patients with and without NP with respect to sensory descriptors
3. To evaluate the relation between neuropathic pain (NP) descriptors and functional status

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with AS according to the Modified NewYork Criteria
* Visual Analogue Scale spinal pain score ≥ 3

Exclusion Criteria:

1. Diabetes mellitus, renal insufficiency, hypothyroidism
2. Postherpetic neuralgia, spinal cord compression
3. Being diagnosed as fibromyalgia in the last month or widespread pain indicating fibromyalgia
4. Malignancy
5. Pregnancy
6. Severe cardiac disease
7. In the last three months medical treatment leading to neuropathy (colchicine etc.)
8. In the last three months drug use for the treatment of fibromyalgia, depression or anxiety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AS patients suffering from spinal pain with severity of 3 or more on 10 cm VAS
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain | Once, at baseline
  It will be assessed using the painDETECT questionnaire. This questionnaire, contains nine questions all of which are selfreport. Seven items are rated on a six point Likert scale and thus are scored between 0-5. These seven questions query some sensations such as burning, tingling or prickling, allodynia, numbness etc. Apart from these seven items, one item assesses the radiation of pain and the other one item looks for the temporal characteristics of pain. A total score of 12 or less indicates neuropathic component is unlikely, 13-18 means possible neuropathic component and 19 or greater means a neuropathic component is likely. Beside these, there are three items in a separate section measuring severity of pain at the time of evaluation, on average and maximum over the past month. This section is not taken into account in scoring.
Neuropathic pain descriptors | Once, at baseline
  In the painDETECT questionnaire, seven items querying sensory abnormalities are scored between 0-5. Each of these abnormal sensations represent a pain descriptor. These descriptors are; burning, tingling, allodynia, pain attacks, thermal hyperalgesia, numbness and pressure hyperalgesia. A descriptor will accepted as positive if it is scored between 3 to 5

SECONDARY OUTCOMES:
Functional status | Once, at baseline
  To measure functional status of patients, Bath Ankylosing Spondylitis Functional Index will be used. It is a 10 item questionnaire querying patients' ability in performing daily activities (such as dressing, bending forward, climbing stairs, reaching a shelf, etc.) on a line of 10 centimeters. The final score is the average of the items, between 0 (no limitation) to 10 (maximal limitation in function).

CONTACTS AND LOCATIONS:
Overall Officials: Taciser Kaya, Prof., MD, Principal Investigator — Izmir Bozyaka Training and Reseach Hospital
Locations (1):
- Izmir Bozyaka Training and Reseach Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi JH, Lee SH, Kim HR, Lee KA. Association of neuropathic-like pain characteristics with clinical and radiographic features in patients with ankylosing spondylitis. Clin Rheumatol. 2018 Nov;37(11):3077-3086. doi: 10.1007/s10067-018-4125-z. Epub 2018 Apr 30. PMID 29713968
- [Background] Bidad K, Gracey E, Hemington KS, Mapplebeck JCS, Davis KD, Inman RD. Pain in ankylosing spondylitis: a neuro-immune collaboration. Nat Rev Rheumatol. 2017 Jul;13(7):410-420. doi: 10.1038/nrrheum.2017.92. Epub 2017 Jun 15. PMID 28615730
- [Background] Heraughty M, Ridehalgh C. Sensory descriptors which identify neuropathic pain mechanisms in low back pain: a systematic review. Curr Med Res Opin. 2020 Oct;36(10):1695-1706. doi: 10.1080/03007995.2020.1790349. Epub 2020 Aug 4. PMID 32609541
- [Background] Ji Y, He Y, Nian X, Sun E, Li L. Inflammatory or Neuropathic Pain: Characteristics and Their Relationships with Disease Activity and Functional Status in Axial Spondyloarthritis Patients. Pain Med. 2019 May 1;20(5):882-888. doi: 10.1093/pm/pny138. PMID 30020521